CLINICAL TRIAL: NCT05382975
Title: A Comprehensive Trauma-sensitive Approach to Physical Activity Promotion in Schools (CSPAP-T)
Acronym: CSPAP-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Pooja Tandon, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003419
Record Dates: First submitted 2022-04-28; First posted 2022-05-19 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Schools will be randomized to start the intervention at different time points
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wedge 1 includes Schools 1 and 2. (Other)
  Interventions: Behavioral: CSPAP-T
- Wedge 2 includes Schools 3, 4, and 5. (Other)
  Interventions: Behavioral: CSPAP-T
- Wedge 3 includes Schools 6, 7, and 8. (Other)
  Interventions: Behavioral: CSPAP-T

INTERVENTIONS:
Behavioral: CSPAP-T — Trauma-adapted CSPAP delivery:
  * Staffing support
  * Trauma-sensitive professional development for teachers and staff
  * Setting specific needs assessment and action planning

SUMMARY:
Investigators will conduct a hybrid implementation-effectiveness trial of a trauma-adapted Comprehensive School Physical Activity Program (CSPAP) intervention. A clustered stepped wedge design will be used, with the duration of the trial being 3 years.

DETAILED DESCRIPTION:
The Comprehensive School Physical Activity Program (CSPAP) is a multi-component approach by which schools use all opportunities for students to be physically active in 5 domains: physical education; physical activity during school; physical activity before and after school; staff involvement; and family and community engagement. Overall, CSPAP-based interventions have had small effect sizes in impacting youth PA, with larger effect sizes seen when more CSPAP domains are included. CSPAP-based interventions are the least effective, and have the most barriers to implementation and sustainability, in school districts that serve a student population that experience intersecting forms of disadvantage and discrimination. Core reasons for this include: (1) youth who have experienced trauma may have unique needs in PA settings, (2) Teachers/staff are not trained to meet the needs of youth who have experienced trauma in PA settings, and (3) staffing constrains the ability of schools to implement new opportunities for PA.

The effectiveness and implementation of a flexible, systems-level intervention to increase opportunities for trauma-sensitive PA in middle schools will be studied. The intervention seeks to support middle schools in increasing opportunities for trauma-sensitive PA practices in all CSPAP domains-addressing two core systems-level barriers to such implementation (staffing and teacher/staff training) and building in flexibility for setting-specific needs assessment and action planning. Core components include (1) provision of a dedicated staff member (via Americorps) to support school PA (via direct staffing and capacity building), (2) setting-specific needs assessment and action planning, and (3) professional development opportunities for teachers, staff, and coaches related to the provision of trauma-sensitive PA.

The study will use a stepped wedge design with a total of 8 middle schools, in which each school will be randomized to start the intervention at different time points. All schools will provide baseline data and will later switch to the intervention phase in random order and in 3 waves. Based on feasibility considerations, 2 schools will switch from control phase to intervention phase in wedge 1, 3 schools will be in wedge 2, and 3 schools will be in wedge 3. Each 2-year intervention phase will be followed by a year when data will be collected to assess sustainability of the intervention. In total, there will be 20 control phase data collections, 24 intervention phase data collections, and 16 data collections during maintenance phase, for a total of 1800 student-assessments (across all schools and all time periods for 20 control and 40 intervention or post-intervention periods). This study will:

1. Assess how intervention exposure is associated with student (accelerometer-measured) PA
2. Assess how intervention exposure is associated with student internalizing and externalizing symptoms and resilient psychosocial function functioning
3. Assess how intervention exposure is associated with change in PA opportunities at the school level
4. Explore systems-level barriers and facilitators to successful intervention implementation and maintenance.

ELIGIBILITY:
Adolescent Inclusion Criteria:

* Age 11-14 (inclusive)
* Attend one of the participating schools during the study period

Teacher/Staff Inclusion Criteria:

* Age 18 or older
* Work at one of the participating schools during the study period

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity - Accelerometer measured. | 2 times per year (Fall, Spring) up to 3 years
  This is the primary outcome for this study and will be collected from a gender stratified random subset of at least 45 students per school, at each time point. Physical activity will be objectively measured using the ActiGraph GT3X worn at the hip for 7 day periods (x 24 hour wear) at each of the data collection timepoints (i.e., fall and spring of each school year).
Change in Internalizing and Externalizing Symptoms. | 2 times per year (Fall, Spring) up to 3 years
  Mental health symptomatology will be measured using the Strengths and Difficulties Questionnaire (self-report version for 11-16 year olds), a brief behavioral screening questionnaire. Scores will be calculated for internalizing problems (emotional+peer symptoms, 10 items, scale 0-20) and externalizing problems (conduct+hyperactivity symptoms, 10 items, scale 0-20). This will be asked in surveys digitally distributed to all students in the fall and spring of each school year. Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Resilient psychosocial functioning | 2 times per year (Fall, Spring) up to 3 years
  Psychological aspects of adolescent resilience will be measured using the 21-item Adolescent Resilience Scale. This three-factor scale measures emotional regulation, positive future orientation, and novelty seeking. This will be asked in surveys digitally distributed to all students in the fall and spring of each school year.

OTHER OUTCOMES:
School-level physical activity | 2 times per year (Fall, Spring) up to 3 years
  The SOPLAY (System of Observing Play and Leisure Activity in Youth) is a validated observation tool designed to obtain observational data on the number of students, their physical activity levels in a specified area (target area) where physical activity could occur, and the predominant type of activity. Data collection will occur for 3 days at each time point, at each school during data collection periods (i.e., fall and spring of each school year) to assess proportion of children engaging in moderate to vigorous physical activity in the various target areas.
School-level physical activity practices. | 2 times per year (Fall, Spring) up to 3 years
  School administrators will complete the Comprehensive School Physical Activity Program Questionnaire (CSPAP-Q) to measure school-level physical activity practices.
School level trauma-sensitive practices | 2 times per year (Fall, Spring) up to 3 years
  School administrators will complete the Trauma Responsive School Implementation Assessment to assess the implementation of trauma-sensitive practices at the school

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States